CLINICAL TRIAL: NCT03579030
Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of RTA 1701 in Healthy Adults
Brief Title: Safety and PK/PD of RTA 1701 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1701-C-1802
Record Dates: First submitted 2018-05-25; First posted 2018-07-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: RTA 1701; RTA 1701 capsules
MeSH Terms: interventions — ORF 50 transactivator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Dose of RTA 1701 or Placebo (Experimental): RTA 1701 capsules or placebo taken orally in a single dose.
  Group 1: RTA 1701 10 mg or matching placebo Group 2: RTA 1701 ≤ 20 mg or matching placebo Group 3: RTA 1701 ≤ 40 mg or matching placebo Group 4: RTA 1701 ≤ 80 mg or matching placebo Group 5: RTA 1701 ≤ 160 mg or matching placebo Group 6: RTA 1701 ≤ 320 mg or matching placebo Group 7: RTA 1701 ≤ 640 mg or matching placebo
  Interventions: Drug: Placebo oral capsule; Drug: RTA 1701 capsules
- Multiple Dose of RTA 1701 or Placebo (Experimental): RTA 1701 capsules, Dose TBD mg or placebo taken orally once daily for 14 weeks.
  Group 8: RTA 1701 ≤40 mg or matching placebo Group 9: RTA 1701 ≤160 mg or matching placebo Group 10: RTA 1701 ≤640 mg or matching placebo
  Interventions: Drug: Placebo oral capsule; Drug: RTA 1701 capsules

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo capsule matched to an RTA 1701 capsule
Drug: RTA 1701 capsules — Capsule containing RTA 1701, multiple dosages

SUMMARY:
This first-in-human, Phase 1, single-center study will evaluate single ascending doses (SAD) and multiple ascending doses (MAD) of RTA 1701 conducted in 2 parts. Part 1 (SAD) of this study will be conducted in approximately 56 healthy participants in up to 7 groups. Each group will consist of up to 8 participants who will be randomized in a 3:1 ratio to receive a single dose of RTA 1701 or placebo, respectively. Safety, tolerability, and available pharmacokinetics in each group will be assessed by the Safety Monitoring Committee prior to dose escalation.

Part 2 (MAD) of this study will be conducted in approximately 30 healthy participants in up to 3 groups and will commence after safety data for the highest dose in the SAD phase has been evaluated. Each group will consist of up to 10 participants who will be randomized in a 4:1 ratio to receive 14 daily doses of RTA 1701 or placebo, respectively. Safety, tolerability, and available pharmacokinetics will be assessed in each dosing group prior to dose escalation

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age is between 18 and 55 years, inclusive;
* Female participants of childbearing potential must:
* Not be pregnant, or lactating, or planning a pregnancy, and
* Be willing to use contraception (hormonal contraceptives, diaphragm, or intrauterine contraception) or abstain from sexual activity (if this is the preferred lifestyle for the participant) for the duration of the study (from initial study drug administration through 90 days after administration of the last dose of study drug);
* Females must have negative results for pregnancy tests performed:
* At screening based on a serum sample, and
* Prior to dosing on Day -1 based on a urine sample;
* If male, participant must be surgically sterile or practice specified methods of contraception from initial study drug administration through 90 days after administration of the last dose of study drug. Male participants must also use a condom during sex to protect male or female partners of male participants from exposure to study drug. In addition to use of a condom, male participants with female partners must also use one of the following acceptable forms of contraception:
* Have had a vasectomy (at least 6 months earlier);
* Partner use of hormonal contraceptives (oral, parenteral, vaginal, or transdermal) for at least 3 months prior to study drug administration;
* Partner use of an intrauterine device;
* Complete abstinence from sexual intercourse (if this is the preferred lifestyle for the participant);
* If male, participant agrees to abstain from sperm donation from initial study drug administration through 90 days after administration of the last dose of study drug;
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 31.0 kg/m2, inclusive;
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG), as judged by the investigator;
* Must voluntarily sign and date each informed consent, approved by a Human Research Ethics Committee (HREC), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* History of clinically significant drug allergies, including allergies to any of the components of the investigational product and/or clinically significant food allergies as determined by the investigator;
* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the investigator;
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines;
* Requirement for any over-the-counter and/or prescription medication, vitamins, and/or herbal supplements on an ongoing basis;
* Use of any OTC medications (over-the-counter), including herbal products, within 7 days prior to Day 1, other than limited paracetamol use (≤ 2 g/day) or oral contraceptive pill. Use of any prescription medication within 14 days or 5 half-lives (whichever is longer), prior to study drug administration, unless in the opinion of the Principal Investigator and/or Medical Monitor the medication will not compromise participant safety or interfere with study procedures or data validity;
* Recent (6-month) history of drug or alcohol abuse;
* Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab) at screening;
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration;
* Receipt of any investigational product within a time period equal to 10 half-lives of the product, if known, or a minimum of 30 days prior to study drug administration;
* Positive screen results for drugs of abuse, alcohol, or cotinine at screening or Day -1;
* Consumption of alcohol within 72 hours prior to study drug administration;
* Consumption of grapefruit, grapefruit products, star fruit, star fruit products, or Seville oranges within the 72-hour period prior to study drug administration;
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration;
* Current enrollment in another clinical study;
* Screening laboratory analyses that show any of the following abnormal laboratory results:
* Alanine transaminase (ALT) level above 1.5 times the upper limit of normal (ULN);
* Aspartate transaminase (AST) level above 1.5 times the ULN;
* Any other laboratory results that are outside of the laboratory normal reference range and considered clinically significant by the investigator;
* Clinically-significant abnormal ECG; ECG with QTc using Fridericia's correction formula (QTcF) > 450 msec (for males) or >460 msec (for females) is exclusionary;
* Consideration by the investigator, for any reason, that the participant is an unsuitable candidate to receive RTA 1701.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 3 weeks
  Safety will be assessed based on the number of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/